CLINICAL TRIAL: NCT06380283
Title: The Feasibility and Clinical Utility of the Use of Virtual Reality for the Management of Pediatric Dental Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Beatriz Ferraz dos Santos, Pediatric dentist; research director, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-10221
Record Dates: First submitted 2024-04-15; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-12

CONDITIONS: Children, Only; Dental Anxiety; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric dental treatment using VR (Experimental): At the beginning of the dental visit, subjects enrolled in the virtual reality (VR) group (n=64) will receive instructions about how to operate the VR system. The research team will then properly fit VR headset onto the child's head and ensure that there are no discomforts. Then, the research team will monitor the intervention using the tablet interface, allowing them to start, pause, and stop the VR intervention. The child will be given 5 minutes to get used to the device. During this time, any adjustments to the headset will be made. The VR intervention will last the duration of the dental procedure, unless told otherwise by the patient, their parent/legal-guardian, or the research team. The entire VR intervention will be closely monitored for any adverse events. Time of play and the patients' compliance of using VR will be noted.
  Interventions: Device: Virtual reality headset
- Control group (No Intervention): Subjects enrolled in the control group (n=64) will receive their dental care using the behavior management techniques recommended by the American Academy of Pediatric Dentistry (i.e., tell-show-so, communicative guidance, distraction through stories and positive reinforcement).

INTERVENTIONS:
Device: Virtual reality headset — Use of a virtual reality headset during pediatric dental care
  Arms: Pediatric dental treatment using VR

SUMMARY:
The use of virtual reality (VR) in pediatric healthcare settings helps to reduce children's pain and anxiety. However, this technology has not been used consistently in pediatric dentistry. Consequently, the goal of this study is to investigate the effectiveness of using a Virtual Reality headset as a distraction technique during dental procedures in children and identify patient and clinician's opinions regarding its use.

This study incorporates a single-site, randomized clinical trial design with two paralleled study groups. One group will receive dental treatment following regular standard of care of behavior management while the second group will receive dental treatment using a Virtual Reality distraction headset. Patients in both groups will complete a questionnaire to assess their perception of pain and anxiety before and after the intervention, as well as their satisfaction with the dental treatment. The dentist providing the treatment will also report their observations relating to patient behavior during dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 and 12 years and their accompanying parent/legal-guardian.
* Children scheduled for one of the following procedures: restorative treatments (amalgam, composite or stainless-steel crowns), pulp therapy and extractions
* Children that can understand and speak French or English.

Exclusion Criteria:

* Children diagnosed with a cognitive, auditory, or cognitive impairment preventing them from interacting with the VR game.
* Children diagnosed with epilepsy or any other condition preventing them from playing the VR game.
* Children requiring urgent dental care
* Children requiring dental treatment with conscious sedation (i.e. nitrous oxide inhalation and/or oral sedation with benzodiazepines)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Children's pain perception during dental treatment | Baseline
  Children's perception of pain during dental treatment will be assessed by the Wong- Baker FACES scale. The 'Face, Legs, Activity, Cry, Consolability' (FLACC), a common behavioral pain external observation scale, will also be used. Higher the score more discomfort and pain experienced by the patient.
Children's fear during dental treatment | Baseline
  The Child Fear Scale will be used to assess the anxiety felt by the participants during dental treatment

SECONDARY OUTCOMES:
Children's acceptability of virtual reality intervention during dental care | Baseline
  The Patient Perception 5-item questionnaire will be used to assess participants acceptability of the VR intervention.
Oral health care provider's acceptability of virtual reality during dental care | Baseline
  A 4-point Likert-scale questionnaire will be used to assess oral health care providers' acceptability of VR during dental treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Dentistry, Montreal Children's Hospital, McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No